CLINICAL TRIAL: NCT05664152
Title: An Open-label, Bridging Study to Assess the Safety and Immunogenicity of BARYCELA Inj. (Live Attenuated Varicella Vaccine for Injection) in Healthy Vietnamese Children Aged Between 12 Months to 12 Years
Brief Title: An Open-label, Bridging Study of BARYCELA Inj. in Healthy Vietnamese Children Aged Between 12 Months to 12 Years
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: GC Biopharma Corp (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: MG1111_VAR_P0302
Record Dates: First submitted 2022-12-02; First posted 2022-12-23 (Actual); Last update posted 2022-12-23 (Actual); Status verified 2022-12

CONDITIONS: Varicella Zoster Virus Infection
Keywords: MG1111; Varicella
MeSH Terms: conditions — Varicella Zoster Virus Infection; Chickenpox

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- MG1111 (Experimental): Participants will be administered subcutaneously with a single dose(0.5 mL dose) of the BARYCELA inj.(MG1111) on the upper arm (brachia lateral).
  Interventions: Biological: MG1111

INTERVENTIONS:
Biological: MG1111 — BARYCELA inj.

SUMMARY:
The goal of this bridging study is to assess the safety and immunogenicity of BARYCELA inj. in healthy Vietnamese children aged between 12 months to 12 years. The main questions it aims to answer are:

* Safety of BARYCELA inj. (Live attenuated varicella vaccine for injection)
* Immunogenicity of BARYCELA inj. (Live attenuated varicella vaccine for injection)

Participants will be administered subcutaneously with a single dose(0.5 mL dose) of the BARYCELA inj.(MG1111) on the upper arm (brachia lateral).

ELIGIBILITY:
Inclusion Criteria:

1. Healthy children aged 12 months to 12 years (inclusive)
2. Subject parent/legal representative willing to provide written informed consent and able to comply with the requirements for the study - Subject able to attend all scheduled visits and to comply with all study procedures
3. Negative history of Varicella and varicella vaccine
4. Subject in good health, based on medical history and physical examination
5. Having a readily identifiable place of residence in the study area, being available for the duration of trial participation, with means of telephone contact.

Exclusion Criteria:

1. Subjects who have a history of Varicella or administration of varicella vaccine
2. Subjects who have hypersensitivity reactions to the component of this Investigational Product, such as gelatin
3. Subjects with untreated active tuberculosis
4. Subjects with a history of Guillain-Barre syndrome
5. Subjects who had received salicylates (aspirin, bismuth subsalicylates) within 4 weeks before administration of investigational product or those who are planning to receive salicylates within 42 days after administration of investigational drug.
6. Subjects who administered anti-viral drug within 4 weeks before administration of investigational product or those who are planning to receive anti-viral drug within 42 days after administration of investigational drug.
7. Subjects who have had an acute febrile episode (at least 38.00C) at some time during the 72 hours before administration of investigational product or those who had any symptom suspected to be allergy including systemic rash.
8. Currently receiving or received any investigational intervention within 30 days prior to the vaccination of study vaccine.
9. Subjects who have completed vaccinations within 4 weeks before enrolment or who are planning to administer other vaccines within 42 days after administration of investigational product.
10. Administered any blood product or intravenous immunoglobulin administration within 44 weeks prior to the vaccination of study intervention
11. Currently receiving or anticipate to receive concomitant immunosuppressive or immune-modifying therapy (excluding inhaled, topical skin and/or eye drop-containing corticosteroids, low-dose methotrexate, or < 2 weeks of daily receipt of prednisone less than 20 mg for subjects who weight more than 10kg and less than 2mg/kg/day for subjects who weight less than 10kg, or equivalent) within 12 weeks prior to the vaccination of study vaccine.
12. Immunosuppressive illness or immunodeficient state, including hematologic malignancy, history of solid organ, bone marrow transplantation, or asplenia.
13. Subject with a history of hypersensitivity to any vaccine or a history of allergic disease or reactions likely to be exacerbated by any component of the study vaccine.
14. Subjects with a severe chronic disease or other clinically significant medical or psychological condition who are considered by the Investigator to be ineligible for the study.
15. Subjects who are pregnant or lactating at the day of screening.
16. Subjects who are planned to participate in another clinical trial during the present trial period.

Ages: 12 Months to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 250 (Estimated)
Dates: Start 2023-02 (Estimated); Primary Completion 2023-04 (Estimated); Study Completion 2023-06 (Estimated)

PRIMARY OUTCOMES:
Safety of BARYCELA inj.: Solicited local and systemic reactogenicity | within 30-minute post vaccination
  The incidence and severity of immediate solicited local and systemic reactogenicity
Safety of BARYCELA inj.: The incidence and severity of solicited local and systemic AEs | during 7 days post vaccination
  The incidence and severity of solicited local and systemic AEs
Safety of BARYCELA inj.: Incidence and severity of unsolicited AEs | during 42 days post vaccination
  The incidence and severity of unsolicited AEs
Safety of BARYCELA inj.: Incidence of adverse event of special interest | during 42 days post vaccination
  The incidence of AE of Special Interest (AESI): varicella-like rash.
Safety of BARYCELA inj.: Vital signs | Day0(Pre vaccination), 42 days post vaccination
  Vital signs
Safety of BARYCELA inj.: Body temperature | Day0(Pre vaccination), 42 days post vaccination
  Body temperature; measured according to standard of care and thermometer instructions.
Safety of BARYCELA inj.: Complete physical examination | Day0(Pre vaccination), 42 days post vaccination
  Complete physical examination; performed at Screening/Enrollment (Day 0) and Final Visit(Day 42).
Safety of BARYCELA inj.: Symptom-directed physical examination | Day0(Pre vaccination), during 42 days post vaccination
  Symptom-directed physical examination (if any symptoms); performed at other timepoints as indicated to assess changes from Screening

SECONDARY OUTCOMES:
Immunogenicity of BARYCELA inj.: Geometric Mean Titer (GMT) | Prior to IP administration and 42 days post vaccination
  Geometric Mean Titer (GMT) of antibody titer measured with gpELISA
Immunogenicity of BARYCELA inj.: Geometric Mean Fold Rise (GMFR) | Prior to IP administration and 42 days post vaccination
  Geometric Mean Fold Rise (GMFR)